CLINICAL TRIAL: NCT04003116
Title: Randomized Clinical Trial to Evaluate the Efficacy and Safety of the Treatment With Supplementary Oxygen in Patients With Intermediate-Risk Pulmonary Embolism (PE)
Brief Title: Air Versus Oxygen for Intermediate-Risk Pulmonary Embolism (AIRE)
Acronym: AIRE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ministry of Health, Spain (Other Government)
Collaborators: Sociedad Española de Neumología y Cirugía Torácica (Other)
Responsible Party: Principal Investigator, David Jimenez, Pulmonary physician, Ministry of Health, Spain
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-000266-37
Record Dates: First submitted 2019-06-27; First posted 2019-07-01 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism | interventions — nitrox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplementary oxygen (Experimental): Supplementary oxygen added to conventional anticoagulant treatment.
  Interventions: Drug: Oxygen gas
- Standard medical therapy (No Intervention): Standard management.

INTERVENTIONS:
Drug: Oxygen gas — Supplementary oxygen during the first 48 hours added to conventional anticoagulant treatment. Patients will receive anticoagulant treatment according to updated guidelines.
  Arms: Supplementary oxygen

SUMMARY:
The primary objective is to evaluate the efficacy of the treatment with supplementary oxygen added to conventional anticoagulant treatment in patients with Intermediate-risk pulmonary embolism.

The secondary objective is to evaluate the safety of the treatment with supplementary oxygen added to conventional anticoagulant treatment in patients with Intermediate-risk pulmonary embolism.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed PE by multidetector computed tomographic pulmonary angiography (MDCT).
* Disfunction of right ventricle (RV to left ventricle [LV] diameter ratio >1.0 in the apical 4-chamber view) in the echocardiogram performed in the first 12 hours after PE diagnosis.
* Signed and dated informed consent of the subject.

Exclusion Criteria:

* <18 years old.
* Allergy to iodinated contrast.
* Renal failure defined as a creatinine clearance less than 30 mL/min, according to the Cockcroft-Gault formula.
* Use of chronic oxygen therapy.
* Hypercapnia (pCO2 >50 mmHg at the time of diagnosis).
* Technically inadequate basal echocardiography.
* Contraindication to anticoagulant therapy.
* Symptoms duration >10 days.
* Haemodynamic instability.
* Participation in other clinical trial for PE treatment during the present clinical trial.
* Inability to use mask or nasal prongs.
* Life expectancy less than 90 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-07-11 (Actual); Primary Completion 2022-04-24 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
Normal right ventricle function at 48 hours | 48 hours
  Right ventricle (RV) to left ventricle (LV) diameter ratio equal or less than 1.0 measured 48 hours after initiation of therapy in normotensive patients with intermediate-risk pulmonary embolism (PE).

SECONDARY OUTCOMES:
Modification RV -LV 7 days | 7 days
  Modification of the right ventricle (RV) to the left ventricle (LV) diameter ratio measured 7 days after initiation of therapy in normotensive patients with intermediate-risk pulmonary embolism (PE).

CONTACTS AND LOCATIONS:
Overall Officials: David Jiménez, Study Chair — IRYCIS, Alcala de Henares University
Locations (7):
- Spain (7):
  - Hospital Universitario Araba, Vitoria-Gasteiz, Alava
  - Hospital Galdakao-Usansolo, Galdakao, Vizcaya
  - Hospital Clínic de Barcelona, Barcelona
  - Clínica Universidad de Navarra, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario y Politécnico La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barrios D, Duran D, Rodriguez C, Moises J, Retegui A, Lobo JL, Lopez R, Chasco L, Jara-Palomares L, Muriel A, Otero-Candelera R, Ruiz-Artacho P, Monreal M, Bikdeli B, Jimenez D; Air vs Oxygen for Intermediate-Risk Pulmonary Embolism Investigators. Oxygen Therapy in Patients With Intermediate-Risk Acute Pulmonary Embolism: A Randomized Trial. Chest. 2024 Mar;165(3):673-681. doi: 10.1016/j.chest.2023.09.007. Epub 2023 Sep 16. PMID 37717936